CLINICAL TRIAL: NCT00191802
Title: Compliance With and Acceptance of Teriparatide Pen Injection in Severely Osteoporotic Patients [CATS]
Brief Title: Compliance and Acceptance of Teriparatide Injection in Severely Osteoporotic Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8370; B3D-CA-GHCP
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Teriparatide

INTERVENTIONS:
Drug: teriparatide

SUMMARY:
The purposes of this study are to evaluate the acceptance of the subcutaneous drug teriparatide over 6 months of therapy in patients with severe osteoporosis in Canada, and to evaluate how often such patients are actually able to use the injection; to obtain additional safety data (side effect data) that will supplement the existing database of adverse events that have been reported to-date in clinical trials by patients treated with teriparatide; to document the prior use of other osteoporosis therapies in this patient population, and ongoing use of other osteoporosis therapies during the study; and to describe the baseline demographics and disease state of these severely osteoporotic patients.The purposes of the study extension are to continue to assess the acceptance of the subcutaneous drug teriparatide over up to 18 months of therapy in patients with severe osteoporosis in Canada, and to continue to assess how often such patients are actually able to use the injection; to obtain additional safety data (side effects) that will supplement the existing database of adverse events that have been reported to date in clinical trials by patients treated with teriparatide.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal woman OR a man at least 30 years of age (who no longer have bone growth)
* In the opinion of the investigator:

  * The patient must have severe osteoporosis (defined as a low bone mass AND a fracture related to osteoporosis), and be at high risk for fracture despite currently available therapies
  * Patients should have failed or been shown to be intolerant to currently commercially available osteoporosis therapies. (Failure of therapy: fracture, or significant loss of bone mass)
  * There should be no other medical causes of the osteoporosis (called idiopathic osteoporosis) except for low estrogen (in women) or low testosterone (in men)
* In the opinion of the investigator, the patient can learn to use the pen type injection delivery system and will be able to use it either alone or with appropriate assistance
* Must be able to understand and sign an approved informed consent document
* Must be able to come in for follow-up visits for the duration of the study.

Exclusion Criteria:

* High blood calcium levels, high parathyroid hormone levels in the blood, high levels of a blood test called alkaline phosphatase that haven't been explained yet.
* Known or suspected bone diseases other than osteoporosis
* Any medical condition that might increase a patient's baseline risk for bone tumors (including prior radiation to the skeleton, Paget's disease, previous bone tumors).
* Recent or currently active kidney stone, OR major problems with kidney function
* Serious ongoing medical problems incompatible with the study (as assessed by the investigator)

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2003-09; Study Completion 2005-10

PRIMARY OUTCOMES:
The primary objective is to determine the acceptance of, and compliance with, 6 months of teriparatide subcutaneous injections in patients with severe osteoporosis who have failed on OR are intolerant to currently available osteoporosis therapies.

SECONDARY OUTCOMES:
To obtain safety data; to document the prior use of other osteoporosis therapies, and concomitant use of other osteoporosis therapies; to describe the baseline demographics and disease state of these severely osteoporotic patients.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9am - 5pm Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (13):
- Canada (13):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Calgary, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Edmonton, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Vancouver, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Winnipeg, Manitoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Moncton, New Brunswick
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, St. John's, Newfoundland and Labrador
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Halifax, Nova Scotia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Hamilton, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, London, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Ottawa, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Toronto, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Montreal, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Saskatoon, Saskatchewan